CLINICAL TRIAL: NCT02469402
Title: Nutritive Efficacy and Safety of a Modified Infant Formula With a Reduced Protein: Content and Improved Protein Quality: LactPro-Minus
Brief Title: Nutritive Efficacy and Safety of a Modified Infant Formula With a Reduced Protein Content and Improved Protein Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Waldkrankenhaus Protestant Hospital, Spandau (Other)
Collaborators: Humana Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Hanna Petersen, Dr. Hanna Petersen, Waldkrankenhaus Protestant Hospital, Spandau
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1026
Record Dates: First submitted 2015-06-09; First posted 2015-06-11 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Overweight
Keywords: reduced; protein; formula; Alpha-lactalbumin; infant
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard infant formula (Active Comparator): Standard infant formula
  Interventions: Dietary Supplement: Standard infant formula
- Protein reduced formula (Experimental): Protein reduced alpha-lactalbumin formula
  Interventions: Dietary Supplement: Protein reduced alpha-lactalbumin formula, with higher levels of alpha-lactalbumin
- Breast-feeding (No Intervention): Exclusive breast-feeding

INTERVENTIONS:
Dietary Supplement: Standard infant formula
  Arms: Standard infant formula
Dietary Supplement: Protein reduced alpha-lactalbumin formula, with higher levels of alpha-lactalbumin
  Arms: Protein reduced formula

SUMMARY:
Formula contains significantly higher total protein concentrations than breast milk. Therefore formula-fed infants have a significantly higher total protein intake in the first few months compared to exclusively breast-fed infants.

The aim is to examine the nutritive efficacy and safety of a modified infant formula with a reduced protein content and improved protein quality in a prospective, double-blind, controled, randomized study. Primary outcome measures are weight gain and growth of young infants under 12 weeks of dietary intake of the new infant formula. Metabolic effects of the qualitative and quantitative changes in the protein content of the new formula will be recorded. Two groups of healthy bottle-fed infants will be compared. The treatment group will be fed for 3 months with an infant formula with decreased protein content. At the same time the protein body of the new formula is modified by enrichment with bovine alpha-lactalbumin.

A control group receives a isocaloric conventional infant formula and a protein body consisting of whey protein and casein in a ratio of 60:40, without specific accumulation of alpha-lactalbumin over the same time-period.

A group of breastmilk fed infants will serve as a reference group. In regular anthropometric controls growth and thriving of the study participants is documented and compared between the different groups.

DETAILED DESCRIPTION:
Breast milk is considered the gold standard for early childhood nutrition, it is optimized in terms of ingredients to the needs of the infant in the first months of life. Formula differ in many ways in their composition to breast milk, e.g. in the structure and concentration of the protein contained.

To ensure adequate supply of the infant with all essential and semi-essential amino acids conventional infant formula contains significantly higher total protein concentrations than breast milk. Therefore formula-fed infants have a significantly higher total protein intake in the first few months compared to exclusively breast-fed infants, and individual amino acids are therefore fed in excess.

The increased intake of protein, and thus the increased intake of some insulinogenic amino acids in infancy (e.g. the branched chain amino acids leucine, isoleucine and valine), is now considered as a possible co-factor for later disposition to overweight and obesity. Breastfeeding induces slower growth of the infant and is proven to be associated with a lower risk of being overweight or obese at the time of school entry (von Kries 1999). The higher protein intake in bottle-fed babies seems to contribute significantly to the differences that can be observed in the growth behavior between breast-fed and bottle-fed children in the first years of life.

Obvious approaches to optimize infant formula are therefore the reduction of protein content, while ensuring an adequate supply of all relevant amino acids similar to breast milk.

Enrichment with alpha-lactalbumin enables the reduction of total protein content in the formula through the qualitative upgrading of the protein body and the high content of essential amino acids, thereby limiting a surplus of protein intake, but at the same time to supply adequate amounts of essential amino acids.

The aim is to examine the nutritive efficacy and safety of a modified infant formula with a reduced protein content and improved protein quality. Primary outcome measures are weight gain and growth of young infants under the 12 weeks of dietary intake of the new infant formula, and metabolic effects of the qualitative and quantitative changes in the protein content of the new formula. Two groups of healthy bottle-fed infants will be compared. The treatment group will be fed for 3 months with an infant formula with decreased protein content. At the same time the body of experimental protein infant formula was modified by enrichment with bovine alpha-lactalbumin.

A control group receives a isocaloric conventional infant formula and a protein body consisting of whey protein and casein in a ratio of 60:40, without specific accumulation of alpha-lactalbumin over the same time period.

A group of breastmilk fed infants will serve as a reference group.

In regular anthropometric controls growth and thriving of the study participants is documented and compared between the different groups. In addition, laboratory tests are carried out, which will examine the influence of diet on insulin response, protein metabolism and specific growth factors.

In a follow-up long-term effects of nutrition on body composition will be recorded by comparing body fat measurements (skinfold thickness-Calipometrie) during the first year of life.

ELIGIBILITY:
Inclusion Criteria:

* At the time of study enrollment apparently healthy newborns / infants without pronounced hyper- or hypotrophy (age-appropriate weight percentiles > 3 and < 97 according to Voigt et al.)
* Maternal decision against breastfeeding (for Formula Groups)

Exclusion Criteria:

* Congenital gastrointestinal malformations, metabolic disease, chromosomal aberration, syndromic disease with significant impact on growth, development, nutrition, immune competence
* Manifestation of a serious disease, which is expected to be accompanied by growth retardation, intestinal transit disruption or the need for special dietary treatment (e.g. hypertrophic pyloric stenosis, cystic fibrosis, Hirschsprung's disease, cow's milk protein intolerance.)
* Decision to administer HA (hypoallergenic) formula due to family atopies (defined by atopic disease of at least one 1 st degree relative: bronchial asthma, atopic dermatitis, pollinosis)
* Participation in another nutritional study

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2014-01; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Composite measure of Growth | 1 year
  height, body weight, head circumference

SECONDARY OUTCOMES:
Daily fluid intake | 3 months
  ml/kg/d

OTHER OUTCOMES:
Plasma concentrations of transthyretin, urea and total protein | 3 months
Body Fat Percentage | 1 year
  skinfold thickness-Calipometrie

CONTACTS AND LOCATIONS:
Overall Officials: Frank Jochum, Dr. med., Principal Investigator — Paul Gerhard Diakonie
Locations (1):
- Evangelisches Waldkrankenhaus Spandau, Berlin, Germany

REFERENCES:
- [Background] von Kries R, Koletzko B, Sauerwald T, von Mutius E, Barnert D, Grunert V, von Voss H. Breast feeding and obesity: cross sectional study. BMJ. 1999 Jul 17;319(7203):147-50. doi: 10.1136/bmj.319.7203.147. PMID 10406746
- [Derived] Gonzalez-Garay AG, Serralde-Zuniga AE, Medina Vera I, Velasco Hidalgo L, Alonso Ocana MV. Higher versus lower protein intake in formula-fed term infants. Cochrane Database Syst Rev. 2023 Nov 6;11(11):CD013758. doi: 10.1002/14651858.CD013758.pub2. PMID 37929831